CLINICAL TRIAL: NCT04816123
Title: The Mass Balance and Biotransformation Study of [14C] Donafenib in Chinese Healthy Adult Male Volunteers
Brief Title: The Mass Balance and Biotransformation of [14C]Donafenib in Healthy Adult Man
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-MB-DNFN-16
Record Dates: First submitted 2021-03-24; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Healthy Male Adult

STUDY DESIGN:
Intervention Model Description: single arm with single dose of 300mg Donafenib, containing about 120μCi [14C]Donafenib
Masking Description: Nonrandomized and open labeled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]Donafenib (Experimental)
  Interventions: Drug: [14C]Donafenib

INTERVENTIONS:
Drug: [14C]Donafenib — Each volunteers received a single 300 mg dose of [14C]donafenib (toluene sulfonic acid) containing a radioactivity dose of 120 μCi as an oral suspension, in fasting within 5 minutes.

SUMMARY:
This study was designed to evaluate the mass balance and biotransformation after single-dose of [14C]Donafenib orally in Chinese healthy adult male volunteers, revealing the overall pharmacokinetic characteristics of Donafenib in humans, and providing a reference for the rational administration.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male adult.
* Age is between 18 and 45, inclusive.
* Body mass index is between 19 and 26, inclusive.
* Voluntarily to provide informed consent form.
* Willing and able to communicate with investigators and complete the trial according to clinical trial protocol.

Exclusion Criteria:

* Any abnormal and clinical significant findings.
* A positive examination result of HBsAg/HBeAg, HIV antibody and treponema pallidum antibody.
* Volunteers who had participated in a radiolabeled clinical study or were exposed to significant levels of radiation for any reasons within the 12 months prior to the study.
* Volunteers who had used of prescription or herbal products that may affect the drug metabolism within 30 days before the study.
* Volunteers who had blood loss/donation up to 400 mL within 3 months before the screening, or received blood transfusion within 1 month.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 6 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
Quantitive analysis of whole radioactivity of excrement of orally administered [14]Donafenib in Chinese healthy adult male volunteers to obtain the mass balance data and the main excretion pathway in human body | from 0 hour to 240 hours after administration
  The percentage of radioactive dose of [14C] radiolabelled Donafenib recovered in urine, faeces and in total
Identification of the main metabolite and biotransformation pathway of Donafenib and investigation of metabolite in plasma by LC-RAM/HRMS | from 0 hour to 240 hours after administration
  Proportion of different metabolites
Quantitive analysis of the concentrations of Donafenib in plasma using the validated LC-MS/MS to obtain pharmacokinetic data | from 0 hour to 240 hours after administration
  The concentrations of Donafenib in plasma

SECONDARY OUTCOMES:
Adverse Events | Up to 7 days (approx) from the start of administration
  Review the relationship between investigational products and all the abnormal and clinically significant findings

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, PhD, Principal Investigator — First Affiliated Hospital of Suzhou Medical College
Locations (1):
- The First Affiliated Hospital of Suzhou University, Suzhou, Jiangsu, China